CLINICAL TRIAL: NCT00221507
Title: Increasing Infant Preventive Health Service Delivery in an Inner City Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Expiration of IRB Approval
Sponsor: University of Colorado, Denver (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-1082; RWJ 048472 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Vaccination; Prevention & Control
MeSH Terms: interventions — Case Management; Patient Navigation

ARMS (4):
- Historical Cohort (No Intervention): This study will first examine risk factors in a defined population of inner city children, using a historical cohort.
- Reminder Recall Outreach (Active Comparator): To determine how well Reminder Recall Outreach will increase immunization rates and well child care delivery in those children most at risk for "falling through the cracks." These studies will be conducted in the Denver Health community health network, the largest integrated community health care system in the United States.
  Interventions: Behavioral: Reminder-Recall-Outreach
- Case Management (Active Comparator): To determine how well Case Management will increase immunization rates and well child care delivery in those children most at risk for "falling through the cracks." These studies will be conducted in the Denver Health community health network, the largest integrated community health care system in the United States.
  Interventions: Behavioral: Case Management
- Patient Navigation (Active Comparator): To determine how well Patient Navigation will increase immunization rates and well child care delivery in those children most at risk for "falling through the cracks." These studies will be conducted in the Denver Health community health network, the largest integrated community health care system in the United States.
  Interventions: Behavioral: Patient Navigator

INTERVENTIONS:
Behavioral: Reminder-Recall-Outreach
  Arms: Reminder Recall Outreach
Behavioral: Case Management
  Arms: Case Management
Behavioral: Patient Navigator
  Arms: Patient Navigation

SUMMARY:
The study hypothesis is that case management using patient navigators ("promatoras" in the Latino community) will increase infant immunization rates and use of well child care in an inner city population of low socioeconomic status.

DETAILED DESCRIPTION:
The overall aim of the proposed project is to increase receipt of a broad array of childhood preventive health services in a population of disadvantaged inner city children. Specific hypotheses concerning risk factors for infant under-immunization and lack of receipt of well child care will be tested. This study will first examine these risk factors in a defined population of inner city children, using a historical cohort. Finally, through the use of a randomized controlled trial in a prospective birth cohort, it will test an intervention, based partly on the evidence gathered from the initial study phases, to increase immunization rates and well child care delivery in those children most at risk for "falling through the cracks." These studies will be conducted in the Denver Health community health network, the largest integrated community health care system in the United States.

Information gathered via rigorous exploration of risk factors for inadequate preventive service receipt in inner city children is especially important at present, because despite rising immunization rates around the country, it is clear that "pockets of need" remain in many urban locations. Children in these pockets of need, in addition to being under-immunized, also are at higher risk for lack of other preventive services, and suffer from higher rates of iron deficiency anemia and lead poisoning. The knowledge gained from both the descriptive and interventional parts of the study will provide crucial information for physicians who care for these children, health care systems that serve them, and policy makers responsible for promoting effective tools and funding their implementation. The information gained herein will also provide important methodological insight for generalists who wish to conduct interventional studies in large urban populations, by further refining existing methods used in design and implementation of large cohort studies in disadvantaged children.

Although this project will be conducted among a population of disadvantaged inner city children, many of the findings from these studies will likely be applicable in health care systems that serve other socioeconomic groups. All primary care physicians who care for children face the challenge of trying to boost childhood immunization rates over 90%, and to increase the delivery of a full spectrum of preventive health services to children. The investigators hope that the evidence from this project will inform and shape both the clinical practice of individual health care providers and health care systems charged with providing preventive health care to children in a wide variety of settings.

ELIGIBILITY:
Inclusion Criteria:

* Any child born at Denver Health Medical Center between 2/1/04 and 1/31/05 who receives primary care at one of 3 community health centers.

Exclusion Criteria:

* No medical care in the Denver Health community health system after 42 days of age.
* Birthweight less than 1500 grams.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2004-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in Infant immunization status
Change in Infant well child care status

SECONDARY OUTCOMES:
Change in Health care utilization
Change in Enrollment in health insurance programs
Change in Screening rates for anemia and lead toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hambidge, MD, PhD, Principal Investigator — UCDHSC
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Hambidge SJ, Phibbs SL, Chandramouli V, Fairclough D, Steiner JF. A stepped intervention increases well-child care and immunization rates in a disadvantaged population. Pediatrics. 2009 Aug;124(2):455-64. doi: 10.1542/peds.2008-0446. Epub 2009 Jul 27. PMID 19651574